CLINICAL TRIAL: NCT02504619
Title: Allogeneic Stem Cell Transplantation of CordIn™, Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells, in Patients With Hemoglobinopathies
Brief Title: Allogeneic SCT of CordIn™, in Patients With Hemoglobinopathies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#01.01.030
Record Dates: First submitted 2015-01-21; First posted 2015-07-22 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CordIn (Experimental): Transplantation of CordIn
  Interventions: Biological: CordIn

INTERVENTIONS:
Biological: CordIn — CordIn™ is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells.

SUMMARY:
CordIn™ is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells. The overall study objectives are to evaluate the safety and efficacy of CordIn™.

DETAILED DESCRIPTION:
CordIn™ is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells.

The trial ends when the last patient completes their last visit. The overall study objectives are to evaluate the safety and efficacy of CordIn™: single ex-vivo expanded cord blood unit transplantation in patients with hemoglobinopathies (sickle cell disease or thalassemia major) following a preparative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for allogeneic SCT for treatment of SCD or thalassemia
* Patients must have one partially HLA-matched CBUs
* Adequate Karnofsky Performance score or Lansky Play-Performance scale
* Sufficient physiological reserves
* Signed written informed consent

Exclusion Criteria:

* Prior allogeneic HSCT
* Evidence of HIV infection or HIV positive serology
* Evidence of active Hepatitis B, Hepatitis C or EBV as determined by serology or PCR
* Active or uncontrolled infection
* Pregnancy or lactation

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Hugues Dalle, MD, Principal Investigator — Robert Debre, Paris, France; Franco Locatelli, MD, Principal Investigator — IRCCS Ospedale Pediatrico Bambino Gesu, Rome, Italy; Allistair Abraham, MD, Principal Investigator — Children's National, Washington DC
Locations (3):
- United States (2):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Children's National, Washington D.C., District of Columbia
- Hôpital Robert Debré, Paris, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CordIn
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CordIn
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 2.8 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Acute Toxicity Associated With the Infusion of CordIn, Within 24 Hours Post-infusion.
Description: The number of patients with grade 4 or 5 toxicity were estimated together with 95% confidence limits based on the binomial distribution. The proportion with toxicity grades 1, 2, and 3 was also estimated.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | CordIn
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: The Percentage of Patients With Donor-derived Engraftment at 42 Days Following Transplantation
Description: One hundred percent of patients engrafted by day forty-two post-transplantation with donor-derived cells.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | CordIn
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Percentage of Overall Survival at 365 Days After Transplantation
Description: The percentage of patients alive at one year post-transplant was estimated using the Kaplan-Meier method.
Time Frame: 365 days
Measure: Count of Participants; unit: Participants
Groups:
- CordIn: Transplantation of CordIn CordIn: CordIn™ is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells.
Arm/Group | CordIn
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Arm/Group | CordIn
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CordIn (N=1)
GvHD (Immune system disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CordIn (N=1)
Hypoalbuminemia (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No